CLINICAL TRIAL: NCT07012382
Title: Association Between Single Gene Polymorphism (rs6746030) and the Success Rate of Inferior Alveolar Nerve Block in Patients Undergoing Endodontic Treatment
Brief Title: Single Gene Polymorphism and the Success Rate of Inferior Alveolar Nerve Block
Acronym: SNP&IANB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Dr. Vivek Aggarwal, Professor, Jamia Millia Islamia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: SNP-Proposal-165
Record Dates: First submitted 2025-05-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Pulpitis - Irreversible
Keywords: irreversible pulpitis; Mandibular Molar; SNP

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to two groups based on the outcome of IANB:
  * Group A (Success Group): Patients with negative response to cold testing and no pain during access cavity preparation.
  * Group B (Failure Group): Patients with persistent response to cold testing and/or intraoperative pain despite IANB.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinding shall be ensured
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Failed inferior alveolar nerve block (Active Comparator): Patients with persistent response to cold testing and/or intraoperative pain despite inferior alveolar nerve block
  Interventions: Procedure: Inferior Alveolar Nerve Block
- Successful inferior alveolar nerve block (Experimental): Patients with negative response to cold testing and no pain during access cavity preparation
  Interventions: Procedure: Inferior-Alveolar-Nerve-Block

INTERVENTIONS:
Procedure: Inferior Alveolar Nerve Block — Administration of standard IANB with 2% lidocaine containing 1:80,000 epinephrine
  Arms: Failed inferior alveolar nerve block
Procedure: Inferior-Alveolar-Nerve-Block — Administration of IANB with 2% lidocaine containing 1:80,000 epinephrine
  Arms: Successful inferior alveolar nerve block

SUMMARY:
The inferior alveolar nerve block (IANB) is one of the most commonly used techniques in dentistry to achieve mandibular anesthesia during endodontic treatment. Despite its widespread use, the success rate of IANB is highly variable, with failure rates reported to range from 30% to 80% in patients with irreversible pulpitis. While several anatomical and clinical factors have been implicated, genetic variations in pain signaling pathways have been increasingly recognized as potential contributors to anesthetic failure. The SCN9A gene, which encodes the voltage-gated sodium channel Nav1.7, plays a critical role in nociception and pain modulation. The single nucleotide polymorphism (SNP) rs6746030 (G>A) in SCN9A has been shown to alter channel function and has been associated with variable pain sensitivity and response to analgesia. This study aims to investigate the association between the SCN9A rs6746030 polymorphism and the success rate of IANB in patients undergoing root canal treatment. A total of 200 patients diagnosed with irreversible pulpitis in mandibular molars will be recruited. Based on anesthetic outcome, they will be divided into two groups: 100 patients with successful IANB and 100 patients with documented anesthetic failure. Buccal swab samples will be collected from each participant, and DNA will be extracted and genotyped using a TaqMan SNP assay. The frequency of SCN9A genotypes (GG, GA, AA) will be compared between the two groups to determine whether there is a statistically significant association with anesthetic outcome. The findings of this study will help identify genetic predictors of anesthetic failure and may provide a foundation for personalized anesthetic strategies in endodontic practice.

DETAILED DESCRIPTION:
The successful administration of local anesthesia is critical for the effective management of pain in endodontic procedures. Among the various local anesthesia techniques, the inferior alveolar nerve block (IANB) is most commonly employed for procedures involving mandibular teeth. However, the IANB often fails to provide profound pulpal anesthesia, especially in cases of irreversible pulpitis. Studies have reported IANB failure rates ranging from 30% to as high as 80% despite proper technique and appropriate choice of anesthetic agents. These failures not only lead to intraoperative pain and patient discomfort but also challenge the clinician's ability to perform the procedure efficiently.Several contributing factors have been proposed to explain this high failure rate, including anatomical variability, inflammation-induced changes in local tissue pH, central sensitization, and psychological factors. More recently, there has been growing interest in the role of genetic predisposition in modulating an individual's response to local anesthetics. Pharmacogenetic studies have suggested that genetic variability in sodium channel genes may influence nociceptive transmission and anesthetic response. The SCN9A gene, located on chromosome 2q24.3, encodes the Nav1.7 voltage-gated sodium channel, which is predominantly expressed in nociceptive neurons of the dorsal root ganglia and trigeminal ganglia (Dib-Hajj et al., 2007). This channel plays a pivotal role in the generation and propagation of action potentials in response to painful stimuli. Mutations and polymorphisms in SCN9A have been linked to various pain syndromes, such as primary erythromelalgia and paroxysmal extreme pain disorder, as well as congenital insensitivity to pain. Notably, the rs6746030 (G>A) SNP, resulting in a missense mutation (R1150W), has been associated with increased pain sensitivity in healthy individuals and altered response to analgesics.

Given this background, it is plausible that genetic variability in SCN9A may also influence the success of local anesthetic techniques like IANB. The proposed study aims to examine whether the SCN9A rs6746030 polymorphism affects the success rate of IANB in patients undergoing root canal treatment for mandibular molars with irreversible pulpitis. Identifying such a genetic association could lead to the development of predictive models for anesthetic response and open avenues for personalized dental anesthesia.

Aims and Objectives: To investigate the association between the SCN9A rs6746030 polymorphism and the clinical success of the inferior alveolar nerve block in patients undergoing endodontic treatment.

This is a prospective case-control genetic association study.A total of 200 patients presenting to the Department of Conservative Dentistry and Endodontics with a diagnosis of irreversible pulpitis in mandibular molars will be enrolled. Participants will be allocated to two groups based on the outcome of IANB:

* Group A (Success Group): Patients with negative response to cold testing and no pain during access cavity preparation.
* Group B (Failure Group): Patients with persistent response to cold testing and/or intraoperative pain despite IANB.

After clinical grouping, a buccal swab will be collected from each participant using sterile DNA collection swabs. The inner cheek will be rubbed for 30-60 seconds, and samples will be stored in sterile tubes at -20°C until processing. DNA will be extracted using the QIAamp DNA Mini Kit (Qiagen, Germany) following the manufacturer's protocol. DNA concentration and purity will be assessed using a NanoDrop spectrophotometer. The rs6746030 SNP in SCN9A will be genotyped using a TaqMan SNP Genotyping Assay (Thermo Fisher Scientific, Assay ID: C_29995789_10). The PCR reactions will be performed in a 96-well format using Applied Biosystems StepOnePlus real-time PCR system. The reaction mix will include TaqMan Genotyping Master Mix, allele-specific probes, and extracted DNA. The thermal profile will consist of an initial denaturation at 95°C for 10 minutes, followed by 40 cycles of denaturation at 95°C for 15 seconds and annealing/extension at 60°C for 1 minute.

Genotype Classification

* GG - Homozygous wild-type.
* GA - Heterozygous.
* AA - Homozygous mutant.

Descriptive statistics will be used to report allele and genotype frequencies. The Hardy-Weinberg equilibrium (HWE) will be assessed using the chi-square test. The association between genotype and anesthetic outcome will be analyzed using chi-square or Fisher's exact test as appropriate. Logistic regression analysis will be used to adjust for confounding factors such as age, gender, and preoperative pain intensity. A p-value of <0.05 will be considered statistically significant. Data will be analyzed using SPSS v25.0 (IBM Corp., USA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years.
* Requiring root canal treatment in mandibular first or second molars diagnosed with irreversible pulpitis.
* Administration of standard IANB with 2% lidocaine containing 1:80,000 epinephrine.
* Ability to provide informed consent.

Exclusion Criteria:

* Systemic conditions affecting pain perception (e.g., diabetes, neuropathies).
* Known allergy to local anesthetics.
* Use of analgesics or anti-inflammatory medications within 24 hours before the procedure.
* Pregnant or lactating women.
* Patients with extensive periapical pathology or swelling.
* Inability to comply with study requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
rs6746030 SNP in SCN9A genotyping | At day 1, at baseline
  The rs6746030 SNP in SCN9A will be genotyped using a TaqMan SNP Genotyping Assay (Thermo Fisher Scientific, Assay ID: C_29995789_10). The PCR reactions will be performed in a 96-well format using Applied Biosystems StepOnePlus real-time PCR system. The reaction mix will include TaqMan Genotyping Master Mix, allele-specific probes, and extracted DNA. The thermal profile will consist of an initial denaturation at 95°C for 10 minutes, followed by 40 cycles of denaturation at 95°C for 15 seconds and annealing/extension at 60°C for 1 minute.
  Genotype Classification
  * GG - Homozygous wild-type.
  * GA - Heterozygous.
  * AA - Homozygous mutant.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Aggarwal, MDS, Principal Investigator — Jamia Millia Islamia
Locations (1):
- Faculty of Dentistry, Jamia Millia Islamia, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD available. The description of the variables, and type of data collected for each individual will be provided on request to the researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 1 month of publication
Access Criteria: The description of the variables, and type of data collected for each individual will be provided on request to the researchers.

REFERENCES:
- [Result] Reimann F, Cox JJ, Belfer I, Diatchenko L, Zaykin DV, McHale DP, Drenth JP, Dai F, Wheeler J, Sanders F, Wood L, Wu TX, Karppinen J, Nikolajsen L, Mannikko M, Max MB, Kiselycznyk C, Poddar M, Te Morsche RH, Smith S, Gibson D, Kelempisioti A, Maixner W, Gribble FM, Woods CG. Pain perception is altered by a nucleotide polymorphism in SCN9A. Proc Natl Acad Sci U S A. 2010 Mar 16;107(11):5148-53. doi: 10.1073/pnas.0913181107. Epub 2010 Mar 8. PMID 20212137
- [Result] Dib-Hajj SD, Yang Y, Black JA, Waxman SG. The Na(V)1.7 sodium channel: from molecule to man. Nat Rev Neurosci. 2013 Jan;14(1):49-62. doi: 10.1038/nrn3404. Epub 2012 Dec 12. PMID 23232607